CLINICAL TRIAL: NCT02288533
Title: Transcranial Direct Current Stimulation (tDCS) Effects in Patients With Chronic Consciousness Disorders
Brief Title: Transcranial Direct Current Stimulation Effects in Patients With Chronic Consciousness Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Sofia Straudi, MD, MD, University Hospital of Ferrara
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Regionale WP2
Record Dates: First submitted 2014-01-16; First posted 2014-11-11 (Estimated); Last update posted 2017-02-03 (Estimated); Status verified 2017-02

CONDITIONS: Minimally Conscious State; TBI
Keywords: Minimally Conscious State; tDCS
MeSH Terms: conditions — Persistent Vegetative State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- real-tDCS (Experimental): Participants will receive tDCS over the primary motor cortex bilaterally (M1). The excitability-enhancing anode electrode (saline-soaked sponge electrode - 16cm2) will be placed over the primary motor cortex, C3 and C4 (10/20 international EEG system). The excitability-diminishing cathode electrode will be placed over the supraorbital area. We will use the following stimulation parameters: intensity of 2 milliampere and for 40 minutes (10 consecutive sessions).
  Interventions: Device: real-tDCS

INTERVENTIONS:
Device: real-tDCS — Participants will receive tDCS over the primary motor cortex bilaterally (M1). The excitability-enhancing anode electrode (saline-soaked sponge electrode - 16cm2) will be placed over the primary motor cortex, C3 and C4 (10/20 international EEG system). The excitability-diminishing cathode electrode will be placed over the supraorbital area. We will use the following stimulation parameters: intensity of 2 milliampere and for 40 minutes (10 consecutive sessions).

SUMMARY:
Chronic consciousness disorders have high level of impact on public health and its costs.

DETAILED DESCRIPTION:
Consciousness disorders have high impact on society and national health system. One of these disorders is vegetative condition in which, as in coma, there isn't any self or environmental consciousness but there is alertness, whereas in minimal state of consciousness at least part of awareness is conserved.

In Emilia Romagna region about 80 people per million of inhabitants are hospitalized after cerebral damage, and after discharge about 1/5 of patients are stabilized in a consciousness disorder.

The diagnosis of these disorders is based on neurobehavioural tests, for example JFK Coma Recovery Scale Revised (CRS-R).

In these patients recovery of state of consciousness is one of the main challenges. There are very little evidences about treatment, it has been proposed the use of therapies that could modulate central nervous system activity, like specific drugs, neuroimaging and neuromodulation techniques such as transcranial magnetic stimulation and repetitive transcranial current stimulation.

A non invasive neuromodulation technique is transcranial direct current stimulation (tDCS) which can modulate cortical excitability: cathodic current reduces excitability whereas anodic current increases it.

In conclusion, tDCS is an easy technique to use, it's not invasive and it's an efficient tool for the modulation of cortical excitability that demonstrated reliable results in healthy subjects.

As the tDCS can modulate cortical excitability it is likely that the combination of this stimulation tool with transcranial magnetic stimulation for the registration of cortical excitability could give important information about cerebral damage in patients with consciousness disorders and to test new treatments. It is also likely that the modification of cortical excitability could induce neurobehavioural changes.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged >18 years old and <70 years old
* diagnosis of disorders of consciousness classified as MCS according to criteria of American Academy of Neurology1.
* traumatic etiology (>12 months after the acute injury)

Exclusion Criteria:

* contraindications to single pulse TMS (TMS will be used to measure cortical excitability) such as metal head implants, history of seizures, metal in the head, implanted brain medical devices.
* contraindications to tDCS such as metal in the head, implanted brain medical devices.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-09; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Coma Recovery Scale Revised (CRS-R) | Change measures (weeks: -2,0,1,2,4)
  behavioural scale (visual, auditory, motor, verbal, communication, arousal)

SECONDARY OUTCOMES:
single-pulse transcranial magnetic stimulation (TMS) | Change measures (weeks: -2,0,1,2,4)
  cortical excitability measures
functional near infrared spectroscopy (fNIRS) | Change measures (weeks: -2,0,1,2,4)
  cerebral perfusion
electroencephalography (EEG) | Change measures (weeks: -2,0,1,2,4)
  To assess if, after tDCS administration, MCS patients could show: electroencephalographic pattern modifications
Circulating Biomarkers | Change measures (weeks: -2,0,1,2,4)
  blood biomarker levels modifications

CONTACTS AND LOCATIONS:
Overall Officials: Sofia Straudi, MD, Principal Investigator — Ferrara Rehabilitation Hospital
Locations (1):
- Ferrara University Hospital, Ferrara, Italy, Italy

IPD SHARING:
Plan to Share IPD: No